CLINICAL TRIAL: NCT03477864
Title: R2810-ONC-16XX: A Phase 1 Neoadjuvant Study of Stereotactic Body Radiation Therapy With Systemic REGN2810 and Intraprostatic Ipilimumab, Alone or in Combination, in Patients With Locally Advanced Prostate Cancer Prior to Radical Prostatectomy
Brief Title: Stereotactic Body Radiation Therapy With REGN2810 and/or Ipilimumab Before Surgery in Treating Participants With Progressive Advanced or Oligometastatic Prostate Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was not accruing
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: Prostate Cancer Foundation (Other); Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 17G.508; JT 10817 (Other: JeffTrial Number)
Record Dates: First submitted 2018-03-19; First posted 2018-03-26 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Stage III Prostate Cancer; Stage IIIA Prostate Cancer; Stage IIIB Prostate Cancer; Stage IIIC Prostate Cancer; Stage IV Prostate Cancer; Stage IVA Prostate Cancer; Stage IVB Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Ipilimumab; CTLA-4 Antigen; Radiosurgery; cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (REGN2810, SBRT, surgery) (Experimental): Participants receive anti-PD-1 monoclonal antibody REGN2810 IV over 30 minutes on day 1 of week 1 and in week 4, and undergo SBRT for 4 fractions on days 2-5 of week 3. Within 14-21 days, participants undergo radical prostatectomy.
  Interventions: Radiation: Stereotactic Body Radiation Therapy (SBRT); Procedure: Radical Prostatectomy; Biological: Anti-PD-1 Monoclonal Antibody REGN2810
- Arm B (ipilimumab, SBRT, surgery) (Experimental): Participants receive ipilimumab via intraprostatic injection on day 1 of week 1, and undergo SBRT for 4 fractions on days 2-5 of week 3. Within 14-21 days, participants undergo radical prostatectomy.
  Interventions: Biological: Ipilimumab; Radiation: Stereotactic Body Radiation Therapy (SBRT); Procedure: Radical Prostatectomy
- Arm C (REGN2810, ipilimumab, SBRT, surgery) (Experimental): Participants receive anti-PD-1 monoclonal antibody REGN2810 as in Arm A and ipilimumab as in Arm B. Participants also undergo SBRT for 4 fractions on days 2-5 of week 3. Within 14-21 days, participants undergo radical prostatectomy.
  Interventions: Biological: Ipilimumab; Radiation: Stereotactic Body Radiation Therapy (SBRT); Procedure: Radical Prostatectomy; Biological: Anti-PD-1 Monoclonal Antibody REGN2810

INTERVENTIONS:
Biological: Ipilimumab — Given via intraprostatic injection
  Other Names: 477202-00-9; 720801; Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; Yervoy; MDX-CTLA4; MDX-010
  Arms: Arm B (ipilimumab, SBRT, surgery); Arm C (REGN2810, ipilimumab, SBRT, surgery)
Radiation: Stereotactic Body Radiation Therapy (SBRT) — Undergo SBRT
Procedure: Radical Prostatectomy — Undergo radical prostatectomy
  Other Names: Prostatovesiculectomy
Biological: Anti-PD-1 Monoclonal Antibody REGN2810 — Given IV
  Arms: Arm A (REGN2810, SBRT, surgery); Arm C (REGN2810, ipilimumab, SBRT, surgery)

SUMMARY:
This phase I trial studies the side effects of anti-PD-1 monoclonal antibody REGN2810 (REGN2810) and/or ipilimumab when given together with stereotactic body radiation therapy before surgery in treating participants with prostate cancer that is growing, spreading, or getting worse, and has spread to other places in the body, or formed a small number of new tumors in one or two other parts of the body. Monoclonal antibodies, such as anti-PD-1 monoclonal antibody REGN2810 and ipilimumab, may interfere with the ability of tumor cells to grow and spread. Stereotactic body radiation therapy is a specialized radiation therapy that sends x-rays directly to the tumor using smaller doses over several days and may cause less damage to normal tissue. Giving anti-PD-1 monoclonal antibody REGN2810 and ipilimumab with stereotactic body radiation therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and tolerability for an established effective dose of systemic REGN2810 and intraprostatic ipilimumab with stereotactic body radiation therapy (SBRT) in patients with locally advanced prostate cancer with or without oligometastatic disease.

SECONDARY OBJECTIVES:

I. To determine overall pathologic response rate after radical prostatectomy. II. To determine prostate-specific antigen (PSA) progression free survival in men treated with REGN2810 and intraprostatic ipilimumab with SBRT.

III. To determine radiographic progression free survival in men treated with REGN2810 and intraprostatic ipilimumab with SBRT.

IV. Acute and chronic adverse events (AEs).

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent for the trial
* Have progressive advanced prostate cancer based on at least one of the following criteria:

  * Gleason score of ≥ 7
  * Any PSA
  * TNM clinical stage T3-T4, N1
* Oligometastatic prostate cancer patients who have not received primary therapy are eligible; (oligometastatic disease is defined as a patient with ≤ 3 metastatic bone lesions on the bone scan or tissue metastasis)
* To be scheduled for a Radical Prostatectomy
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale
* Absolute neutrophil count (ANC) ≥ 1000 /mcL within 7 days of treatment initiation
* Platelets ≥ 150,000 / mcL within 7 days of treatment initiation
* Hemoglobin ≥ 9 g/dL or ≥ 5.6 mmol/L within 7 days of treatment initiation
* Lymphocytes ≥ 500 / mcL within 7 days of treatment initiation
* Serum creatinine ≤ 1.5 X upper limit of normal (ULN) OR measured or calculated creatinine clearance (CrCl) ≥ 50 mL/min for subject with creatinine levels > 1.5 X institutional ULN within 7 days of treatment initiation

  * Glomerular filtration rate (GFR) can also be used in place of creatinine or CrCl
* Serum total bilirubin ≤ 1.5 X ULN within 7 days of treatment initiation

  * Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN within 7 days of treatment initiation
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) ≤ 2.5 X ULN within 7 days of treatment initiation
* International normalized ratio (INR) or prothrombin time (PT) ≤ 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or INR is within therapeutic range of intended use of anticoagulants within 7 days of treatment initiation
* Activated partial thromboplastin time (aPTT) ≤ 1.5 X ULN unless subject is receiving anticoagulant therapy as long as aPTT is within therapeutic range of intended within 7 days of treatment initiation

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent within 4 weeks of the first dose of treatment
* Prior treatment with an agent that blocks PD-1/PD-L1 pathway or other immune modulating agents within fewer than 4 weeks of 4 half-lives
* Has a diagnosis of immunodeficiency or is receiving any systemic steroid therapy or any form of immunosuppressive therapy within 7 days prior to day 1 of trial treatment
* Has had a prior monoclonal antibody within 4 weeks prior to study day 1 or who has not recovered (i.e., ≤ grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
* Has had prior treatment with idelalisib
* Has had prior or current treatment with Androgen Deprivation Therapy
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., ≤ grade 1 or at baseline) from adverse events due to a previously administered agent

  * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
  * Note: Subjects with ≤ grade 2 neuropathy are an exception to this criterion and may qualify for the study
* Has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial urothelial cancer, or superficial bladder cancer that has undergone potentially curative therapy
* Has an active autoimmune disease requiring systemic treatment within the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs) or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents
* Has evidence of interstitial lung disease, active, non-infectious pneumonitis
* Has evidence of significant liver disease
* Has an active infection requiring systemic therapy; prior to dosing with REGN2810 the subject must be at least 5 half-lives from their last dose of antibiotic
* Has a history of listeriosis or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Has a contraindication to administration of amoxicillin, ampicillin, ciprofloxacin, erythromycin, gentamycin, penicillin, trimethoprim/sulfamethoxazole, and vancomycin
* Is expecting to spontaneously conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment
* Has contraindication to administration of non-steroidal anti-inflammatory drugs (NSAIDS)
* Is or has an immediate family member (spouse or children) who is investigational site or staff directly involved with this trial, unless prospective Institutional Review Board (IRB) approval (by chair or designee) is given allowing exception to this criterion for a specific subject

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12-24 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2019-11-04 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events as defined by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 criteria | Up to 70 days
  Will be assessed by quantifying the toxicities and grades 3 and 4 experienced by subjects who have received REGN2810 + ipilimumab in combination with radiation therapy, including serious adverse events (SAEs) and events of clinical interest (ECIs). Time-to-event continual reassessment (TITE-CRM) design will be used to confirm the safety of the treatments based on toxicities.

SECONDARY OUTCOMES:
Overall pathologic response rate | Up to 2 years
  Will be presented with appropriate confidence intervals (95%, unless otherwise specified).
Prostate specific antigen (PSA) progression free survival | Up to 2 years
  Will be estimated using the Kaplan-Meier method.
Radiographic progression free survival | Up to 2 years
  Will be estimated using the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Dicker, MD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/